CLINICAL TRIAL: NCT05166044
Title: Safety Observation of Enterovirus 71 Inactivated Vaccine (Vero Cell) Combined Immunization With Other Vaccines in Shanghai
Brief Title: Safety Observation of Enterovirus 71 Inactivated Vaccine (Vero Cell) Combined Immunization in Shanghai
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: EV71-SH-2020-01
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2021-12

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — This study did not involve sample collection.Only adverse reactions/events at 3 days, 14 days and 30 days after vaccination of EV71 vaccine and the other vaccine were collected by face-to-face or telephone follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Safety group: All of the participants(N=12500) received one dose of EV71 vaccine and one of other vaccines(such as MMR vaccine,encephalitis vaccine,mumps vaccine,inactivated poliomyelitis vaccine,influenza vaccine and so on ) at the same time.
  Interventions: Biological: EV71 Inactivated Vaccine

INTERVENTIONS:
Biological: EV71 Inactivated Vaccine — The EV71 vaccine was manufactured by Sinovac Biotech Co,And inactivated EV71 virus antigen was no less than 3.0EU in 0.5 mL of aluminium hydroxide solution per injection.

SUMMARY:
This study is an open clinical trial of the EV71 vaccine (Vero cell), Inactivated manufactured by Sinovac Research & Development Co.,Ltd.The purpose of this study is to evaluate the safety of EV71 vaccine (Vero cell), Inactivated co-administration with other vaccines

DETAILED DESCRIPTION:
This study is an open clinical trial in children aged 6-71 months old. The purpose of this study is to evaluate the safety of EV71 vaccine (Vero cell), inactivated co-administration with other vaccines.The EV71 vaccine was manufactured by Sinovac Biotech Co.A total of 12500 subjects aged 6-71 months old were enrolled.All subjects received one dose of EV71 vaccine and one of other vaccines(such as MMR vaccine,encephalitis vaccine,mumps vaccine,inactivated poliomyelitis vaccine,influenza vaccine and so on ) at the same time.

ELIGIBILITY:
Inclusion Criteria:

* 6 months ≤ Age of enrollment ≤71 months;
* Voluntary and self-funded completion of EV71 vaccine combined immunization with one of the other type I or II vaccines;
* The subject and/or guardian can understand and voluntarily sign the informed consent form;
* Subjects and their legal guardians are able to attend follow-up visits and follow all study procedures (such as cooperating in completing safety observation notes).

Exclusion Criteria:

-

Ages: 6 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In this study,only children aged 6-71 months old who were judged by vaccination doctors to be eligible for vaccination and voluntary and self-funded completion of EV71 vaccine combined immunization with one of the other type I or II vaccines were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Safety index-incidence of local and systemic adverse reactions | From 0 to 3 days after vaccination
  Incidence of local and systemic adverse reactions 0 to 3 days after each dose of EV71 vaccine combined immunization with other vaccines (except live attenuated vaccines)
Safety index-the incidence of local and systemic adverse reactions | From 0 to 14 days after vaccination
  The incidence of local and systemic adverse reactions 0 to 14 days after each dose of EV71 vaccine combined with live attenuated vaccine
Safety index-The incidence of adverse reactions | From 0 to 30 days after vaccination
  The incidence of adverse reactions 0-30 days after vaccination of EV71 vaccine combined immunization with other vaccines.
Safety index-Incidence of serious adverse reactions | From 0 to 30 days after vaccination
  Incidence of serious adverse reactions 0 to 30 days after vaccination of EV71 vaccine combined immunization with other vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Linlin Wu, Master, Principal Investigator — Shanghai Center for Disease Control and Prevention
Locations (6):
- China (6):
  - Baoshan District Center for Disease Control and Prevention, Baoshan, Shanghai Municipality
  - Jing'an District Center for Disease Control and Prevention, Jing’an, Shanghai Municipality
  - Minhang District Center for Disease Control and Prevention, Minhang, Shanghai Municipality
  - Putuo District Center for Disease Control and Prevention, Putuo, Shanghai Municipality
  - Qingpu District Center for Disease Control and Prevention, Qingpu, Shanghai Municipality
  - Xuhui District Center for Disease Control and Prevention, Xuhui, Shanghai Municipality